CLINICAL TRIAL: NCT02830282
Title: Surveillance Markers of Utility for Recurrence After Neoadjuvant Chemotherapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 16113
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Blood Collection

SUMMARY:
This is a nested multicenter, prospective cohort study within the I-SPY 2 TRIAL for women undergoing neoadjuvant chemotherapy for primary breast cancer who are also undergoing definitive surgical resection and have clinical or radiographic evidence of residual tumor at the completion of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment on the treatment phase of the I-SPY 2 TRIAL
* Completed a standard neoadjuvant chemotherapy regimen or assigned treatment on I-SPY 2 and planning definitive surgical resection. Participants who have discontinued assigned treatment on I-SPY 2, switched to standard of care, and have completed a standard neoadjuvant chemotherapy regimen are still considered eligible.
* Pre-surgical imaging or clinical examination demonstrating residual disease in the breast. Participants with any extent of enhancement attributable to tumor on the pre-surgical MRI are eligible. No minimum extent of palpable tumor pre-surgery is required.
* Willing to undergo bone marrow aspiration and blood specimen collection per protocol specifications
* No clinical evidence of distant metastatic disease. Pre-chemotherapy staging scans are sufficient in the absence of any symptoms or subsequent clinical evidence suggesting distant metastases
* Age 18 or over and are able to give informed consent

Exclusion Criteria:

* Individuals under the age of 18
* Individuals who cannot understand and give informed consent. We will not be assessing decisional capacity; determination of ability to give informed consent will be at the discretion of the treating physician.
* Pregnancy. Participants in the parent I-SPY 2 TRIAL are screened for pregnancy at enrollment and pregnancy is an exclusion criteria. No additional screening for pregnancy is required for participants enrolling on SURMOUNT. However if a study participant does become pregnant while on study or during the course of the 10 year follow-up, the study participant will remain on the study protocol and will not be withdrawn. Because this is an observational study and does not have a therapeutic component, there will be no increased risk to following a study participant through annual blood draws and medical information abstraction from the medical chart who may or may not become pregnant during the course of the follow-up period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women undergoing neoadjuvant chemotherapy for primary breast cancer who are undergoing definitive surgical resection and have clinical or radiographic evidence of residual tumor at the completion of chemotherapy
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-07; Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Number of disseminated tumor cells (DTCs), | 2 years
Number of circulating tumor cells (CTCs) | 2 years
Number of other circulating tumor biomarkers (CBMs) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela DeMichele, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States